CLINICAL TRIAL: NCT04225390
Title: A Phase 2, Single Arm Study on Dacarbazine (DTIC) Followed by Immunotherapy Re-challenge in Unresectable or Metastatic Melanoma With Primary Resistance to PD-1/PD-L1 or PD-1 + CTLA-4 Blockade
Brief Title: Preconditioning of Tumor, Tumor Microenvironment and the Immune System to Immunotherapy
Acronym: PROMIT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Collaborators: University Hospital Regensburg (Other); Wuerzburg University Hospital (Other); Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PROMIT
Record Dates: First submitted 2020-01-03; First posted 2020-01-13 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-01

CONDITIONS: Immunotherapy
Keywords: immune checkpoint blockade; resistance; dacarbazine
MeSH Terms: interventions — Dacarbazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Dacarbazine (Experimental): Dacarbazine (day1 and day21) 850 mg/m² i.v. followed by re-exposure to the previous immunotherapy
  Interventions: Drug: Dacarbazine (DTIC)

INTERVENTIONS:
Drug: Dacarbazine (DTIC) — Dacarbazine powder for IV solution
  Other Names: DTIC

SUMMARY:
PROMIT is a single arm phase 2 trial evaluating the clinical activity of immune checkpoint blockade (ICB) after administration of dacarbazine (DTIC) in patients with unresectable or metastatic, BRAF wildtype melanoma with primary resistance to anti-programmed-cell-death-1 (PD-1/PD-L1) or PD-1 plus anti-cytotoxic-T-lymphocyte antigen 4 (CTLA-4) blockade therapy. If the activity is clinically meaningful, DTIC could become a new therapeutic option to break primary resistance to immunotherapy.

DETAILED DESCRIPTION:
PROMIT is a phase 2, single arm, open label study of DTIC followed by combined immune checkpoint blockade (ICB) therapy or PD-1/PD-L1-blockade monotherapy in adult (≥ 18 years) subjects with previously treated, unresectable or metastatic melanoma (Stage III or Stage IV melanoma as per the AJCC staging system). Subjects must be BRAF wildtype and must have shown primary resistance to ICB. Fresh tumor tissue from an unresectable or metastatic site of disease must be available.

Subjects will be treated with DTIC 850 mg/m² day 1 and 21 i.v. (DTIC phase). Afterwards, patients will receive combined ipilimumab (3 mg/kg) and nivolumab (1 mg/kg) 4 times every 3 weeks i.v. OR nivolumab 240 mg every 2 weeks OR pembrolizumab 200 mg every 3 weeks (ICB re-exposure phase; EMA-approved dosing scheme). By the end of the ICB phase, response will be documented (primary endpoint). A safety follow-up for treatment-related adverse events will be performed until 30 days after the last dose of combined ICB. Patients will be followed for survival every 12 weeks after the end of the combined ICB phase (second primary endpoint). Tumor and blood samples will be assessed over the course of the study to evaluate changes in tumor, tumor microenvironment and immune system.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed metastatic melanoma
2. Progression after checkpoint inhibitor therapy (PD-1/PD-L1 or PD-1 + CTLA-4 blockade)
3. Accessible tumor metastases
4. ECOG 0 or 1
5. Adequate organ function

Exclusion Criteria:

1. Uvea melanoma, mucosal melanoma
2. Previous chemotherapy in metastatic disease
3. Previous response to checkpoint inhibitor therapy (PD-1/PD-L1 or PD-1 + CTLA-4 blockade) in metastatic disease
4. BRAF V600 mutation
5. Active brain metastases
6. Autoimmune disease requiring more than 10 mg prednisolone daily or other immunosuppressive drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2020-01-13 (Actual); Primary Completion 2026-01-15 (Actual); Study Completion 2026-01-15 (Actual)

PRIMARY OUTCOMES:
Rate of participents with CR, PR, SD or PD | week 14
  A patient is defined as responder if a complete response (CR) or partial response (PR) can be seen. A patient with stable disease (SD) or progressive disease (PD) will be defined as non-responder.

SECONDARY OUTCOMES:
Overall survival (OS) | up to 5 years
  Overall survival (OS), defined as the time between study inclusion and date of death (any cause). For subjects without documentation of death, OS will be censored on the last date the subject was known to be alive. OS will be followed continuously while subjects are on the study drug and every 12 weeks via phone contact after subjects discontinue the treatment phase.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Erlangen, Bavaria, Germany